CLINICAL TRIAL: NCT04344171
Title: CovidDB: The Covid-19 Inpatient Database
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ClarData (Other)
Responsible Party: Sponsor
Other Study IDs: CovidDB
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Sars-Cov-2; Covid-19; antiviral therapy; ventilation; ECMO
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the project is to better understand the Covid-19 inpatient course of the disease and to quickly identify the positive experiences in the treatment in order to update guidelines for the treatment and use of medication.

DETAILED DESCRIPTION:
The exponentially increasing number of SARS-CoV-2 infected people, despite the influence of the currently existing non-medical measures, is generating a rapidly increasing number of inpatients, some of whom need artificial ventilation. The average focus is on the extent to which the hospitals' capacities will be sufficient to adequately treat all patients. Regardless of this, it can be expected that even if the non-medical measures are successful, the number of inpatients treated will remain high in the course of the pandemic. With regard to the distribution of infection, it can be expected that clinics with a wide range of expertise will have to treat a large number of Covid-19 patients.

So far, however, there is little to no experience in treating patients. In addition to epidemiological data, only case descriptions and some Chinese studies mostly from Wuhan based on fewer patients are available. In view of the rapidly spreading pandemic, preprints are increasingly being used. What has been missing so far is a uniform, structured recording of the courses of Covid-19 inpatients handled by many clinics, which goes beyond the epidemiological events in terms of depth of detail. With this documentation of real processes, the basis for a large number of studies and the associated better understanding of the disease process could be created.

The current dynamics make it imperative that the clinics, even those who have not received the most up-to-date scientific knowledge, cannot wait for the results of studies, but rather need concrete help in the treatment of patients. Efficient assistance within the framework of a close exchange between the treatment units is only possible with a multicentre, uniform documentation environment.

The aim of the project is to better understand the Covid-19 inpatient course of the disease and to quickly identify the positive experiences in the treatment in order to update guidelines for the treatment and use of medication.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 inpatients

Exclusion Criteria:

* assumed Covid-19 patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is focused on all Covid-19 inpatients which are treated in the recruited hospitals.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Outcome comparison between different antiviral therapies | through study completion, an average of 1 year
  Different antivirals and their combinations will be tested and the outcome (cured/deceased) will be assessed
Outcome comparisons between ventilation types | through study completion, an average of 1 year
  Different ventilation types will be tested and the outcome (cured/deceased) will be assessed
Identification of risk factors | through study completion, an average of 1 year
  Clinical and laboratory risk factors will be recorded and the outcome (cured/deceased) will be assessed
Number of days in hospital vs. clinical classification | through study completion, an average of 1 year
  Correlation between number of days in hospital and worst clinical classification will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Julia Ferencz, MD, Principal Investigator — ClarData; Hans-Rudolf Tinneberg, Prof., Principal Investigator — University of Giessen
Locations (9):
- Germany (8):
  - RoMed - Klinikum Bad Aibling, Bad Aibling
  - DONAUISAR Klinikum Deggendorf, Deggendorf
  - DONAUISAR Klinikum Dingolfing, Dingolfing
  - RoMed - Klinikum Prien am Chiemsee, Prien am Chiemsee
  - RoMed - Klinikum Rosenheim, Rosenheim
  - Universitätsklinikum Ulm, Ulm
  - RoMed - Klinikum Wasserburg Am Inn, Wasserburg am Inn
  - Klinikum Altmühlfranken, Weißenburg
- Timiş County Emergency Clinical Hospital, Timișoara, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Budweiser S, Bas S, Jorres RA, Engelhardt S, von Delius S, Lenherr K, Deerberg-Wittram J, Bauer A. Patients' treatment limitations as predictive factor for mortality in COVID-19: results from hospitalized patients of a hotspot region for SARS-CoV-2 infections. Respir Res. 2021 Jun 4;22(1):168. doi: 10.1186/s12931-021-01756-2. PMID 34098967
- See also: This is the website of the study and database — https://www.covid-db.com